CLINICAL TRIAL: NCT06614439
Title: Proximal Versus Total Gastrectomy for Advanced Proximal Gastric Cancer: A Retrospective Double-Center Propensity Score-Matched Cohort Study
Brief Title: PG Versus TG for Advanced PGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 202408135RIND
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-09

CONDITIONS: Gastric Adenocarcinoma; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal gastrectomy (Experimental)
  Interventions: Procedure: proximal gastrectomy
- Total gastrectomy (Active Comparator)
  Interventions: Procedure: total gastrectomy

INTERVENTIONS:
Procedure: proximal gastrectomy — proximal gastrectomy
  Arms: Proximal gastrectomy
Procedure: total gastrectomy — total gastrectomy
  Arms: Total gastrectomy

SUMMARY:
We conducted a retrospective study on patients with pathological stage II-III PGC who underwent PG or TG from 2013 to 2023. Propensity score-matching was applied to adjust for tumor size and stage between the PG and TG groups at a 1:1 ratio. We evaluated the procedural safety, oncological, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Proximal gastric adenocarcinoma after total or proximal gastrectomy.

Exclusion Criteria:

* Non-curative resections
* Non-adenocarcinoma histology
* Distally located tumors or middle/proximally located tumors for which distal margin could not be secured by PG
* Remnant gastric cancer
* Clinically T1N0 tumors smaller than 3 cm for which PG was clearly indicated

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
five-year overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsin-Chu County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Chae YS, Yun WG, Kim JC, Park JK, Kim MG, Kim J, Cho YS, Kong SH, Park DJ, Lee HJ, Yang HK. Long-Term Outcome of Proximal Gastrectomy for Upper-Third Advanced Gastric and Siewert Type II Esophagogastric Junction Cancer Compared With Total Gastrectomy: A Propensity Score-Matched Analysis. Ann Surg Oncol. 2024 May;31(5):3024-3030. doi: 10.1245/s10434-024-15048-8. Epub 2024 Feb 19. PMID 38372863
- [Background] Peng R, Yue C, Wei W, Zhou B, Wen X, Gu RM, Ming XZ, Li G, Chen HQ, Xu ZK. Proximal gastrectomy may be a reasonable choice for patients with selected proximal advanced gastric cancer: A propensity score-matched analysis. Asian J Surg. 2022 Oct;45(10):1823-1831. doi: 10.1016/j.asjsur.2021.09.029. Epub 2021 Oct 9. PMID 34642056
- [Background] Rosa F, Quero G, Fiorillo C, Bissolati M, Cipollari C, Rausei S, Chiari D, Ruspi L, de Manzoni G, Costamagna G, Doglietto GB, Alfieri S. Total vs proximal gastrectomy for adenocarcinoma of the upper third of the stomach: a propensity-score-matched analysis of a multicenter western experience (On behalf of the Italian Research Group for Gastric Cancer-GIRCG). Gastric Cancer. 2018 Sep;21(5):845-852. doi: 10.1007/s10120-018-0804-3. Epub 2018 Feb 8. PMID 29423892
- [Background] Sugoor P, Shah S, Dusane R, Desouza A, Goel M, Shrikhande SV. Proximal gastrectomy versus total gastrectomy for proximal third gastric cancer: total gastrectomy is not always necessary. Langenbecks Arch Surg. 2016 Aug;401(5):687-97. doi: 10.1007/s00423-016-1422-3. Epub 2016 May 4. PMID 27143021
- [Background] Lee S, Son WJ, Roh YH, Song JH, Park SH, Cho M, Kim YM, Hyung WJ, Kim HI. Indication of Proximal Gastrectomy for Advanced Proximal Gastric Cancer Based on Lymph Node Metastasis at the Distal Part of the Stomach. Ann Surg Open. 2021 Nov 24;2(4):e107. doi: 10.1097/AS9.0000000000000107. eCollection 2021 Dec. PMID 37637877